CLINICAL TRIAL: NCT04135248
Title: A Randomized Control Trial in People With Type 1 Diabetes Mellitus Who Will Fast Ramadan: Does Insulin Timing and Dose Matter?
Brief Title: A Randomized Control Trial in People With Type 1 Diabetes Who Will Fast Ramadan: Does Insulin Timing and Dose Matter?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Other Study IDs: RA HM 2019-017
Record Dates: First submitted 2019-08-25; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Flash Glucose Monitoring, Time-in-Range, Fasting, Ramadan
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IDF-DAR arm: Insulin management according to IDF-DAR guidelines (IDF-DAR arm) during the fasting period.
- DAFNE arm: Insulin management according to local experience (DAFNE arm) during the fasting period.

SUMMARY:
Fasting Ramadan is one of the five pillars of Islam and requested only from healthy adults to abstain from eating and drinking from sunrise to sunset. People with type 1 diabetes mellitus (TIDM) are exempted from fasting, as their chronic condition could be adversely affected by fasting. Nevertheless, many insist on fasting and it has been experienced and advocated that with proper education and follow-up with health care providers, people with uncomplicated T1DM could safely fast Ramadan.

Adopted IDF-DAR guidelines for people with diabetes planning to fast Ramadan are available but are based on opinions and largely untested. These current guidelines recommend a significant reduction in insulin doses and a change of the timing of basal insulin and highlight the increased risk of hypoglycemia. Our local DAFNE patient's experience with fasting during the past years points towards no significant changes in insulin timing with minor reductions of insulin without a significant increase in the risk of hypoglycemia. There is no randomized control trial to test the efficacy of the IDF-DAR guidelines specifically looking at changing basal insulin timing This study aims to assess whether insulin doses require reduction and change of timing during Ramadan. We aim to compare the effectiveness and safety of two management strategies. This will help to provide robust guidelines to help both health care professionals and people with type 1 diabetes

DETAILED DESCRIPTION:
INTRODUCTION/BACKGROUND

Diabetes and Ramadan (DAR) and IDF international collaboration created the IDF-DAR guidelines which include the practical recommendations for HCP to better manage people with diabetes who plan to fast Ramadan. The National Institute for Health and Clinical Excellence has recommended implementation of structured education programs to help individuals enhance their knowledge about diabetes and improve their management techniques. The educational program needs to ensure that patients can cope with specific situations such as exercise, illness which should extend to religious fasting.

We have developed and adopted a 5-day educational program widely used in the UK for delivery in Kuwait. The course trains adults with Type 1 Diabetes in the UK to manage their condition more effectively using multiple injections. As part of our course, DAFNE graduates receive yearly Ramadan diabetes educational specific session (separate from the main 5-day course) and all DAFNE graduates are invited. During the 6 hours session, we seek patients' views, willingness to fast and introduced to the specific food that commonly consumed during Ramadan. Previous personal experiences of fasting and problems encountered are collected. Patients who are intending to fast and whom we deem safe to undertake this, receive clear and practical guidance on safe fasting during Ramadan.

Current Gaps in the Literature

Most intervention studies up to date have been performed in controlled conditions, using a small number of participants and with a short duration of intervention, ie not closely related to real-life. The variability of insulin regimens, dietary patterns and physical activity levels and the complexity of ways in which they are tested make it difficult to identify the individual effects of each component on diabetes outcomes. As a result, further research is needed to help expand the currently available knowledge regarding the management of diabetes and its associated complications when fasting during Ramadan. We believe that large, randomized, controlled intervention trials are necessary to broaden our understanding of the implications of fasting and evaluate guidance without bias. Further research into the effect of fasting during Ramadan on both high (measured by SMBG and HbA1C) and low glucose (measured by the incidence of hypoglycemia) is required. Robust evaluation of evidence-based guidelines will lead to useful practical assistance for patients who can fulfill religious obligations despite the additional burden of insulin-treated diabetes. This pilot study builds on an educational program, DAFNE which includes many of the elements of flexible eating and insulin dose adjustment which should permit patients to fast safely.

Study Rationale

Adopted IDF-DAR guidelines are available but recommend a significant reduction in insulin doses and change to the timing of basal insulin for MDI users. There is no evidence that fasting increases the risk of hypoglycemia, and glucose tends to be higher during Ramadan, as a result of a reduction in insulin doses.

Local DAFNE patient's experience with fasting during the past years points towards no significant changes in insulin doses (minor reductions were needed in basal or bolus insulin doses) without the need of the change of basal insulin timing, however we are not aware without running a randomized control trial (RCT) to test DAFNE guidelines versus DAR-IDF guidelines.

OBJECTIVES / HYPOTHESIS

The primary objectives of this study are to assess whether insulin doses require reduction during Ramadan and change of timing and whether fasting increases the risk of hypoglycemia for people with T1DM who fast Ramadan.

Hypothesis:

This study hypothesized no changes in insulin dose timing and fasting does not increase the risk of hypoglycemia.

METHODOLOGY

Potential patients will be identified via DAFNE database at DDI. Candidate subjects who are current users of (FSL) and administer insulin via (MDI) will be contacted by phone and will be offered conditional participation in the study. Those agreeable will be given the consent form with the preferred language (Arabic or English) and will be scheduled a study visit. The same will be done for insulin pump users.

Study design

Open-label randomized controlled trial in people with uncomplicated T1DM fasting during Ramadan (1 month) comparing insulin management according to IDF-DAR guidelines (IDF-DAR arm) and local experience (DAFNE arm), on time spent in range (TIR) of 4-10 mmol/L, and hypoglycaemic self-reported episodes.

Primary outcome:

1. Percentage TIR 4-10mmol/L
2. Rate of self-reported hypoglycemia by participants

Secondary outcomes:

1. Percentage time <4mmol/L
2. Percentage time >10mmol/L
3. Number of sensors detected hypoglycaemic events
4. Number of days needed to break the fast

Inclusion/exclusion criteria:

Mentioned in separate section

Intervention:

The intervention in this study is insulin dosing and timing during Ramadan, and it will be assessed by creating two groups of participants that are similar to one another in all respects, except to the intervention to be assessed. Participants will be DAFNE graduates who were trained properly on carbohydrate counting and adjusting insulin doses according to the carbs consumed. The whole cohort will be using the same insulin regimen; multiple daily injections (MDI) and monitoring glucose using the same monitoring systems; flash glucose monitoring (FGM) system: FreeStlye Libre (FSL) Reader and sensors, and self-monitoring of blood glucose (SMBG) using the FreeStyle optimum test strips, or insulin pump.

The null hypothesis is that there is no difference in the rates of hypoglycemia between basal insulin taken at iftar time versus bedtime in people with T1DM during fasting Ramadan.

Ramadan Workshop

DAFNE structured education program was conducted to all subjects in a stage their life with T1DM. Consequently, subjects are familiar with carbohydrate counting and aware of dose adjustments needed to cover their meals. Nevertheless, this workshop will include food tables with real food models of traditional Ramadan plates. The workshop includes advices on healthy eating habits during Ramadan. General instructions will be provided to all participants which are part of DAFNE Ramadan protocol.

Ramadan Visits, Daily messages, and Calls

Visits: Weekly or whenever required, to upload FSL reader and adjust doses without crossing the arm recommendations for adjustments. This can be done in person or via the cloud Daily Messages: Did you fast full day? If no, was it due to hypoglycemia, and did you check BG to confirm hypoglycemia? Daily count of hypoglycemic episodes? Was all confirmed with SMBG? Are you wearing a glucose sensor, and scanning readings at least once every 8 hours? Calls: If participant was not answering messages, calls will be initiated. A message or call should be performed in the last day of Ramadan to instruct participants about the insulin dosing and timing post-Ramadan

Post-Ramadan Visit:

1. Upload FSL reader
2. Physical examination will be repeated, including weight and routine blood will be collected again including HbA1C, FBC, U&Es with eGFR, full chemistry, urine ACR within three months
3. This will conclude the study visits for the subject

DATA ANALYSIS

For statistical analysis, this can be done using two-tailed unpaired t-test as we are comparing results of different subjects who are in different conditions and the change can be rise or fall in time in range.

Telemonitoring data including daily questionnaires, WhatsApp messages, food logs, and meal pictures will be collected and added to an excel sheet for analysis.

FreeStlye libre software will be used to extract reports and data export readings of FSL readers. The following analysis will be carried out for both arms and for all fasted days:

1. Total average of 24 hours of glucose
2. Estimated A1c
3. Percentage time in range 4.0-10mmol/L
4. Percentage time spent <4.0mmol/L
5. Percentage of time spent >10mmol/L
6. Low glucose events
7. Low glucose duration
8. Total patient-reported hypoglycemia events (from telemonitoring data mentioned above) One-way ANOVA to compare means of percentage time in all above glucose ranges with an alpha <0.05

IMPORTANCE OF THE RESEARCH OUTCOMES

IDF-DAR guidelines recommend reducing insulin doses in people with T1DM or insulin-dependent T2DM to prevent hypoglycemia especially in the 3 to 4 hours before iftar, in addition to changing the basal insulin timing. DAFNE earlier work at DDI demonstrated that fasting Ramadan did not require a significant reduction of background basal insulin (most 5-10% if needed) without reduction of meal bolus insulin. It also advocates that there is no increased risk of hypoglycemia in Ramadan if done with the support of diabetes with prior education and close glucose monitoring. However, there is significant evidence that glucose tends to be higher during Ramadan especially post-iftar, as a result of eating feasting behavior and most probably a reduction in insulin doses as per guidelines. There is no consensus between guidelines and local experience and no evidence about the cut-off reduction in insulin doses which requires running this randomized control trial which hypothesized that the change in eating behavior in Ramadan does not change insulin requirement and carb counting will provide safe insulin dosing during Ramadan similar to that outside Ramadan

ETHICAL CONSIDERATIONS Informed Consent Forms

We will give a patient information sheet for the participant to keep and ask for written informed consent. We will document that 3 copies have been distributed: one to the participant, another to his/her doctor and one for the study team

CONFIDENTIALITY

All hard copies of any study material will be kept in locked cabinets on the premises of DDI. Subject identifiable information will be only available to study team and ethics committee for inspection in case this becomes required.

ELIGIBILITY:
Inclusion Criteria:

1. T1DM for 12 months or more
2. Age >21 years old
3. Current user of FSL and plan to use it during Ramadan
4. HbA1C <10%
5. Planning to fast Ramadan
6. People with T1DM on insulin pump

Exclusion Criteria:

1. Any significant diabetes-related complications including, but not limited to

   1. Any recent episode of severe hypoglycemia in the preceding 12 months
   2. Any recent DKA in the preceding 12 months
   3. Diabetic nephropathy with eGFR <60ml/minute/1.73m2
   4. Diabetic retinopathy ≥R2, ≥M1
   5. Peripheral neuropathy
   6. Active or recent foot ulcers
   7. HbA1c greater than 10%.
2. Hypoglycaemia unawareness
3. Pregnancy or plannig for pregnancy over the duration of the study
4. Breast feeding
5. Active malignancy
6. Uncontrolled thyroid disorders
7. Not able to attend study visits
8. Not able or not willing to give written informed consent
9. Not DAFNE graduates

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes subjects, enrolled in the DAFNE center, Dasman Diabetes Institute, Kuwait.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-04-17 (Estimated)

PRIMARY OUTCOMES:
Percentage time spent in glucose range 4-10mmol/L | 30 days
  FreeStlye libre software will be used to extract reports and data export readings of FSL readers. Data will be collected during the whole month of Ramadan fasting for the outcome measure.
Rate of self-reported hypoglycaemia | 30 days
  The data of self- reported hypoglycaemic episode will be collected daily basis by using telecommunication and whatsapp massage.

SECONDARY OUTCOMES:
Percentage time at the glucose level <4mmol/L or >10mmol/L | 30 days
  The percentage time spent in hypo- and hyperglycemic range will be determined.
Number of days needed to break the fast | 30 days
  All patients will be instructed to break their fast if blood glucose reach 3.9 mmol/L confirmed with SBMG.

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa Al-Ozairi, MBChB(UK), Principal Investigator — Dasman Diabetes Institute, Kuwait
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Dasman, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided